CLINICAL TRIAL: NCT06734117
Title: Clinical Performance of Elecsys® Troponin T hs Gen 6 in Subjects With Symptoms of Acute Coronary Syndrome
Brief Title: A Study of Elecsys® Troponin T hs Gen 6 in Participants With Symptoms of Acute Coronary Syndrome
Acronym: PERFORM-TSIX
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diagnostics GmbH (Industry); Roche Diagnostics Operations, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CIM RD005477
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Signs and Symptoms of Acute Coronary Syndromes: The study population will be a consecutive all-comers cohort consisting of patients with signs and symptoms of acute coronary syndromes presenting to the emergency department. Participants will be diagnosed and treated according to the local standard of care at the study site.
  Interventions: Diagnostic Test: Elecsys® Troponin T hs Gen 6; Procedure: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Elecsys® Troponin T hs Gen 6 — It is an immunoassay for the in vitro quantitative determination of cardiac troponin T (cTnT) in human serum and plasma using cobas e platforms. This investigational immunoassay is intended to aid in the diagnosis of myocardial infarction.
Procedure: Blood sample collection — Blood will be collected from each recruited individual by a healthcare practitioner at five time points after emergency department presentation.

SUMMARY:
This prospective, non-interventional, single arm, longitudinal cohort multicenter study will recruit approximately 5600 consecutive all-comers, consisting of patients with signs and symptoms of acute coronary syndromes (ACS) who present in the emergency department (ED). The main objective of the study is to determine the clinical performance of Elecsys Troponin T hs Gen 6 versus the centrally adjudicated clinical diagnosis at various time points after ED presentation using the previously determined clinical cut-off of a universal 99th percentile upper reference limit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Signed Informed Consent Form
* Troponin or other cardiac marker determination planned as part of suspected acute coronary syndromes routine care
* Demonstrating symptoms suggestive of acute coronary syndrome and/or myocardial ischemia, such as any of the following:

  1. Chest pain, pressure, or a burning sensation across the precordium and epigastrium;
  2. Pain that radiates to neck, shoulder, jaw, back, upper abdomen, or either arm;
  3. Acute onset or worsening dyspnea;
  4. Nausea, vomiting or indigestion;
  5. Lightheadedness or syncope;
  6. Diaphoresis;
  7. Generalized weakness or fatigue; OR, asymptomatic subjects or patients with atypical symptoms in whom myocardial infarction is being suspected.

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 5600 consecutive all-comers with signs and symptoms of acute coronary syndromes presenting to the emergency department.
Sampling Method: Probability Sample
Enrollment: 5429 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Elecsys® Troponin T hs Gen 6 Against the Centrally Adjudicated Clinical Diagnosis at Timepoint T3aid | T3aid (121 to 240 minutes) after participant presentation at the emergency department
  The sensitivity of a diagnostic test is the percentage of true positive (TP) tests out of all patients with a condition. It is calculated as follows: (TP)/(TP + false negatives (FN))*100%.

SECONDARY OUTCOMES:
Sensitivity of Elecsys® Troponin T hs Gen 6 Against the Centrally Adjudicated Clinical Diagnosis at Specified Timepoints | T0aid (0 to 60 minutes), T1aid (61 to 120 minutes), T5aid (241 to 360 minutes), and T6+aid (>360 minutes) after participant presentation at the emergency department
  The sensitivity of a diagnostic test is the percentage of true positive tests out of all patients with a condition. It is calculated as follows: (TP)/(TP + FN)*100%.
Specificity of Elecsys® Troponin T hs Gen 6 Against the Centrally Adjudicated Clinical Diagnosis at Specified Timepoints | T0aid (0 to 60 minutes), T1aid (61 to 120 minutes), T3aid (121 to 240 minutes), T5aid (241 to 360 minutes), and T6+aid (>360 minutes) after participant presentation at the emergency department
  The specificity of a diagnostic test is the percentage of true negative (TN) tests out of all patients who do not have a condition. It is calculated as follows: (TN)/(TN + false positives (FP))*100%.
Negative Predictive Value of Elecsys® Troponin T hs Gen 6 Against the Centrally Adjudicated Clinical Diagnosis at Specified Timepoints | T0aid (0 to 60 minutes), T1aid (61 to 120 minutes), T3aid (121 to 240 minutes), T5aid (241 to 360 minutes), and T6+aid (>360 minutes) after participant presentation at the emergency department
  The negative predictive value of a diagnostic test is the percentage of true negative tests out of all of the negative findings. It is calculated as follows: (TN)/(TN + FN)*100%.
Positive Predictive Value of Elecsys® Troponin T hs Gen 6 Against the Centrally Adjudicated Clinical Diagnosis at Specified Timepoints | T0aid (0 to 60 minutes), T1aid (61 to 120 minutes), T3aid (121 to 240 minutes), T5aid (241 to 360 minutes), and T6+aid (>360 minutes) after participant presentation at the emergency department
  The positive predictive value of a diagnostic test is the percentage of true positive tests out of all of the positive findings. It is calculated as follows: (TP)/(TP + FP)*100%.
Negative Predictive Value of Fast Rule-Out of Myocardial Infarction Using Elecsys® Troponin T hs Gen 6 and the European Society of Cardiology 0/1-Hour Algorithm | T0fast (0 to 60 minutes) after participant presentation at the emergency department and T1fast (30 to 90 minutes from T0fast sample)
  The negative predictive value of a diagnostic test is the percentage of true negative tests out of all of the negative findings. It is calculated as follows: (TN)/(TN + FN)*100%.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- United States (26):
  - El Centro Regional Medical Center, El Centro, California
  - UCSD La Jolla ED, La Jolla, California
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Parkview Research, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Health, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University at Buffalo / Buffalo General Hospital, Buffalo, New York
  - University of Buffalo - Erie County Medical Center, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, High Point Medical Center, High Point, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Health Florence Medical Center, Florence, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Eastside Research Associates, Redmond, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Aspirus Medical Group, Wausau, Wisconsin
- Medical University Vienna, Vienna, Austria
- Bulgaria (2):
  - MHAT "Heart and Brain", Burgas
  - MHAT "Heart and Brain", Pleven
- China (7):
  - Peking University First Hospital, Beijing
  - Dongguan People's Hospital, Dongguan
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Shanghai Tongren Hospital, Shanghai
  - TEDA International Cardiovascular Hospital, Tianjin
  - Tongji Hospital, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
- Germany (3):
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
- Japan (3):
  - Tokyo Bay Urayasu Ichikawa Medical Center, Chiba
  - Kurashiki Central Hospital, Okayama
  - Omihachiman Community Med Center, Ōmihachiman
- Catharina Ziekenhuis, Eindhoven, Netherlands
- Akershus University Hospital (AHUS), Oslo, Norway
- Spain (2):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Alvaro Cunqueiro, Vigo
- Switzerland (2):
  - University Hospital Basel, Basel
  - Luzerner Kantonsspital, Lucerne
- United Kingdom (2):
  - NHS Lothian, Edinburgh
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniels LB, Giannitsis E, Mueller C, Meex SJR, Buehlmann D, Kurtoic D, Bendig G, Cole M, Body R, Christenson RH, Cobbaert C, deFilippi CR, Eggers KM, Inoue K, Jaffe AS, McCarthy CP, McCord J, Neumann JT, Omland T, Papendick C, Sandoval Y, Tan JWC, Than MP, Twerenbold R, Mills NL, Peacock WF; TSIX investigators. Clinical performance of the next generation Elecsys Troponin T high-sensitivity Gen 6 assay in acute coronary syndrome (PERFORM-TSIX): study design. Clin Res Cardiol. 2026 Jan 19. doi: 10.1007/s00392-025-02842-x. Online ahead of print. PMID 41553478